CLINICAL TRIAL: NCT00920543
Title: A Multicenter, Randomized, Double-blind, Parallel Group, 40-week Comparison of Asthma Control Using Bronchial Hyperresponsiveness as an Additional Guide to Long-term Treatment in Adolescents and Adults Receiving Either Fluticasone Propionate/Salmeterol DISKUS Twice Daily or Fluticasone Propionate DISKUS Twice Daily (or Placebo BID if Asymptomatic)
Brief Title: GSK BHR Study (Sont)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM40086
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fluticasone propionate (Active Comparator)
  Interventions: Drug: Placebo; Drug: FP 100mcg; Drug: FP 500mcg; Drug: FP 250mcg
- Fluticasone propionate/salmeterol combination (Active Comparator)
  Interventions: Drug: Placebo; Drug: FSC 100/50mcg; Drug: FSC 250/50mcg; Drug: FSC 500/50mcg

INTERVENTIONS:
Drug: Placebo — Twice daily dosing
Drug: FP 100mcg — Twice daily dosing
  Arms: Fluticasone propionate
Drug: FP 500mcg — Twice daily dosing
  Arms: Fluticasone propionate
Drug: FP 250mcg — Twice daily dosing
  Arms: Fluticasone propionate
Drug: FSC 100/50mcg — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination
Drug: FSC 250/50mcg — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination
Drug: FSC 500/50mcg — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination

SUMMARY:
The purpose of this study was to determine whether asthma control and reduced bronchial hyperresponsiveness could be achieved and maintained at a lower dose of inhaled corticosteroids with ADVAIR DISKUS twice-daily or FP twice-daily in adult and adolescent subjects with persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis
* Controller medications or moderate inhaled corticosteroid dose
* Evidence of reversibility

Exclusion Criteria:

* Life-threatening asthma
* Asthma instability
* Concurrent respiratory disease
* Drug allergy
* Respiratory tract infection
* Systemic corticosteroid use
* Immunosuppressive medication use
* Positive pregnancy test
* Tobacco use
* Site affiliation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2003-02; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Average inhaled corticosteroid treatment dose over the treatment period | Every 8 weeks for the 40 week treatment period

SECONDARY OUTCOMES:
Pulmonary function measures | Every 8 weeks for the 40 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (48):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Petoskey, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Absecon, New Jersey
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Rockville Centre, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Tigard, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Morgantown, West Virginia
- Brazil (2):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, Ponce, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dorinsky P, Yancey S, Baitinger L, Stauffer J. Measuring Airway Hyperresponsiveness: Does it add to routine measures of clinical efficacy in guiding asthma therapy? Eur Respir J 2006;28(50):319s.
- [Background] Kerwin EM, Nathan RA, Meltzer EO, Ortega HG, Yancey SW, Schoaf L, Dorinsky PM. Efficacy and safety of fluticasone propionate/salmeterol 250/50 mcg Diskus administered once daily. Respir Med. 2008 Apr;102(4):495-504. doi: 10.1016/j.rmed.2007.12.002. Epub 2008 Feb 21. PMID 18206361
- [Background] Koenig SM, Murray JJ, Wolfe J, Andersen L, Yancey S, Prillaman B, Stauffer J, Dorinsky P. Does measuring BHR add to guideline derived clinical measures in determining treatment for patients with persistent asthma? Respir Med. 2008 May;102(5):665-73. doi: 10.1016/j.rmed.2007.12.023. Epub 2008 Mar 6. PMID 18328683
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAM40086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register